CLINICAL TRIAL: NCT03452501
Title: An Observational, Prospective Cohort Study to Evaluate the Safety and Effectiveness of Remsima® in the Treatment of Inflammatory Bowel Disease Among Saudi Arabia Patients Diagnosed With Crohn's Disease, Ulcerative Colitis, or Fistulizing CD
Brief Title: Safety and Effectiveness Study of Remsima® in the Treatment of Inflammatory Bowel Diseases Among Saudi Arabia Patients
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RMS-KSA-2016-03
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Fistulizing Crohn's Disease; Ulcerative Colitis
Keywords: Infliximab; Remsima; Biosimilar; Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis; Fistulizing Crohn's Disease; Observational; Follow up; Safety; Effectiveness; Disease modifying anti-rheumatic drugs; Tumor necrosis factor-alpha inhibitors
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; CT-P13

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Naïve group: Newly diagnosed patients
  Interventions: Drug: Infliximab
- Switched group: Patients who received at least one dose of Infliximab reference medicinal product (RMP) before the first infusion of Remsima®
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — A vial containing powder for concentrate for solution for infusion. Each vial contains: Infliximab 100 mg
  Other Names: Remsima®

SUMMARY:
The purpose of this observational study is to assess the safety and effectiveness of biosimilar Infliximab in patients with inflammatory bowel disease (IBD) in Saudi Arabia where no visits or intervention(s) additional to the daily practice will be performed.

DETAILED DESCRIPTION:
A multicenter, observational, prospective, cohort study to assess the safety and effectiveness of biosimilar Infliximab (Remsima®) in newly diagnosed and in switched IBD patients diagnosed with active Crohn's disease (CD), fistulizing CD, or Ulcerative Colitis (UC). Each patient is expected to be treated for a total of 38 weeks if naive or 40 weeks if switched. The study duration will be between 46 and 48 weeks (up to 12 months). Follow-up is expected to end 8 weeks after the last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients with moderate to severe active CD who have not responded despite a full and adequate course of therapy with corticosteroids and/or immunosuppressive agents, or who are intolerant to or have medical contraindications to such therapies.
* Adult patients with fistulizing active CD who have not responded despite a full and adequate course of therapy with conventional treatment (including antibiotics, drainage and immunosuppressive therapy).
* Adult patients with moderate to severe active UC who have had an inadequate response to conventional therapy including corticosteroids and 6-mercaptopurine (6-MP) or azathioprine (AZA), or who are intolerant or have medical contraindications to such therapies.
* Switched patients who received at least one dose of Infliximab reference medicinal product (RMP) before the first infusion of Remsima®.
* Patients who agree to join the study and give a written informed consent

Exclusion Criteria:

* - Patients with a known history of hypersensitivity to infliximab, to other murine proteins, or to any of the excipients (Sucrose, Polysorbate 80, Monobasic sodium phosphate and/or Dibasic sodium phosphate).
* Patients who have shown intolerance or inefficacy to biologics for IBD treatment.
* Female patients who are known to be pregnant or breastfeeding.
* Patients with a past or present history of chronic infection with Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV), or those with positive test at screening.
* Patients who are diagnosed with tuberculosis (TB) or previously diagnosed with TB with no evidence of complete resolution
* Patients with severe or chronic infections (e.g. sepsis, abscesses, opportunistic infections, invasive fungal infections), or severe or chronic infection, without sufficient documentation of complete resolution following treatment
* Patients with recent exposure to persons with active TB, or a positive test result for latent TB at Screening. A patient who has received at least the first 30 days or recommended period of country-specific TB prophylactic therapy and intends to complete the entire course of therapy may be enrolled. Recommended methods to screening latent TB are interferon-γ release assay [IGRA] test, with a chest X-ray, however, other methods could be used according to local guideline.
* Patients with moderate or severe heart failure (New York Heart Association NYHA class III/IV).
* Patients for whom the treatment with Tumor necrosis factor-alpha (TNF-α) blockers is concerning due to a history of malignancy within the previous five years prior to enrollment or a history of herpes zoster within one month prior to enrollment, may be excluded at the investigator's discretion.
* Patients who meet any of the contraindications to the administration of infliximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from approximately 6 sites in Saudi Arabia
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) to Remsima® | 12 months
  Number, type, severity and frequency of adverse events (AEs), serious AEs (SAEs), and clinically relevant changes in laboratory tests (according to laboratory reference ranges), in addition to the incidence of latent tuberculosis (TB) activation (as an adverse event) and the incidence of hepatitis B virus HBV, hepatitis C virus (HCV), and human immunodeficiency virus (HIV) will be assessed

SECONDARY OUTCOMES:
Proportions of naïve patients with CD achieving clinical response or remission based on Crohn's Disease Activity Index (CDAI) | Up to 12 months
  Clinical response is defined by a decrease in CDAI score from baseline of at least 70 points (Response-70). Clinical remission score < 150 for naïve patients with CD
Proportion of switched patients with CD achieving disease control | Up to 12 months
  Disease control is defined as the absence of disease worsening, with worsening defined as increase in CDAI of 70 points or more from the qualifying score with a total score of 175 or more and an increase in CDAI of 35% or more from baseline, or the introduction of a new treatment for active CD
Proportion of naïve patients with fistulizing CD achieving clinical response or remission | Up to 12 months
  Clinical response is defined as reduction of at least 50% from baseline in the number of draining fistulas. Clinical remission is defined as the absence of draining fistulas
Proportion of switched patients with fistulizing CD achieving disease control | Up to 12 months
  Disease control is defined as no loss of response, with loss of response defined as the recrudescence of draining fistulas, the need for a change in medication for CD, the need for additional therapy for persistent or worsening luminal disease activity, the need for a surgical procedure for CD, or the discontinuation of study medication owing to a perceived lack of effectiveness
Proportion of naïve patients with UC achieving clinical response or remission based on Partial Mayo Score and mucosal healing | Up to 12 months
  Clinical response is defined as a decrease in partial Mayo scores from baseline of 2 points or more and 30% or more, with an accompanying decrease in the subscore for rectal bleeding of 1 point or more, or an absolute subscore for rectal bleeding of 0 or 1). Clinical remission is defined as a total partial Mayo score of 2 points or less, with no individual sub-score of more than 1 point), Mucosal healing (assessed through endoscopy, and defined by Mayo endoscopic subscore of 1 point or less)
Proportion of switched patients with UC achieving disease control. | Up to 12 months
  Disease control is defined as the absence of disease worsening, with worsening defined by an increase in partial Mayo score of 3 points or more from baseline [before switching] and a partial Mayo score of 5 points or more).

CONTACTS AND LOCATIONS:
Locations (4):
- Saudi Arabia (4):
  - King Abdulaziz University Hospital, Jeddah
  - Prince Sultan Military Medical City, Riyadh
  - King Abdullah International Medical Research Center, Riyadh
  - King Saud Medical City, Riyadh